CLINICAL TRIAL: NCT03429192
Title: A Multi-centre Real-world Non-interventional Observational Study to Explore Clinical Characteristics of Lymph Skip Metastases and Prognoses of N2 Patients With Non-small Cell Lung Cancer
Brief Title: A Study to Explore Clinical Characteristics and Prognoses of N2 Patients With Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Tianjin Chest Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Lingyu Huang, Professor, Tianjin Chest Hospital
Other Study IDs: TJ-N2LC-01
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Chinese, real-world evidences, NSCLC, lymph skip metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N2 non-small cell lung cancer: Chinese patients with N2 non-small cell lung cancer
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgeries plus dissection of lymph nodes

SUMMARY:
A study to compare patient survivals in the N2 patients with non-small cell lung cancer in the subgroups of lymph skip metastases and non-skip metastases

DETAILED DESCRIPTION:
A multi-centre real-world non-interventional observational study to retrospectively collect the study data on patient demographic/tumor biological characteristics and clinical treatments to compare patient survivals in the N2 patients with non-small cell lung cancer in the subgroups of lymph skip metastases and non-skip metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgeries from 2014 to 2017;
* Pathologically diagnosed patients with non-small cell lung cancer;
* Age > 18 years old;
* Patients with chest surgeries before hospitalization;
* Patients with N2 lymph nodes (+) after surgeries who received lymphadenectomy (Group 10 and 11 lymph nodes);

Exclusion Criteria:

- Patients with radiotherapies, chemotherapies and biological therapies for tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically diagnosed Chinese NSCLC patients with chest surgeries and lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 2653 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Difference in overall survival (OS) | 2014 - 2017
  OS difference in the subgroups of N2 patients with lymph skip metastases and non-skip metastases

SECONDARY OUTCOMES:
Percentage of N2 patients with lymph skip metastases | 2014 - 2017
  Percentage of N2 patients with lymph skip metastases

OTHER OUTCOMES:
Difference in overall survival (OS) (in the subgroups of patients) | 2014 - 2017
  OS difference in subgroups of patients with lymph skip metastases and non-skip metastases categorised by baseline characteristics
Hazard factors of overall survival | 2014 - 2017
  Hazard factors of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xun Zhang, PhD, Principal Investigator — Tianjin Chest Hospital
Locations (9):
- China (9):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China People's Liberation Army Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huaxi Technology University, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Xi'an Tangdu Hospital, Xi'an, Shanghai Municipality
  - Huaxi Hospital Affiliate to Sichuan University, Chengdu, Sichuan
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Li X, Fu X, Liu L, Liu Y, Zhao H, Li Y, Hu J, Xu L, Liu D, Yang H, Zhang X. Survival benefit of skip metastases in surgically resected N2 non-small cell lung cancer: A multicenter observational study of a large cohort of the Chinese patients. Eur J Surg Oncol. 2020 Oct;46(10 Pt A):1874-1881. doi: 10.1016/j.ejso.2019.12.015. Epub 2019 Dec 18. PMID 31902592